CLINICAL TRIAL: NCT01531517
Title: Study of the Efficacy of Topical Application of Royal Jelly and Panthenol (PedyPhar® Ointment) on the Diabetic Foot Ulcers, An Open Label, Randomized, Non-placebo-controlled Study
Brief Title: Study of the Efficacy of PedyPhar® Ointment on the Diabetic Foot Ulcers
Acronym: PED111
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: inability to recruit patients
Sponsor: European Egyptian Pharmaceutical Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pedyphar2012
Record Dates: First submitted 2012-02-06; First posted 2012-02-13 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Diabetic Foot Ulcer
Keywords: Pedyphar; Ointment; Healing; Diabetic; Foot Ulcer
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer | interventions — royal jelly; dexpanthenol; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pedyphar (Experimental): Ointment
  Interventions: Drug: Royal Jelly and Panthenol (PedyPhar® Ointment)
- Panthenol (Active Comparator): Ointment
  Interventions: Drug: Panthenol Ointment

INTERVENTIONS:
Drug: Royal Jelly and Panthenol (PedyPhar® Ointment) — the following will be done to each patient depending on the number of the visit:
  1. Assessment of the patient for inclusion/exclusion criteria
  2. Informed consent process
  3. Medical history of the patient
  4. Blood withdrawn for investigation
  5. Drainage of the ulcer if there is a collection
  6. Revascularization as needed and indicated by APSV done at visit 0.
  7. Swab from the ulcer for culture and micro-organism count: on detailed visits only.
  8. Debridement as needed.
  9. Dressing:
     * Inspection and assessment of the ulcer
     * Irrigation using 500 ml of saline or as required.
     * Drying of the ulcer (leave to dry)
     * Spread a layer of 3 - 5 mm of PedyPhar on a dressing and then apply the dressing to the ulcer
     * Fix the dressing to the ulcer
  Other Names: Pedyphar; Panthenol; Royal Jelly; Ointment; Diabetic Foot Ulcer
  Arms: Pedyphar
Drug: Panthenol Ointment — the following will be done to each patient depending on the number of the visit:
  1. Assessment of the patient for inclusion/exclusion criteria
  2. Informed consent process
  3. Medical history of the patient
  4. Blood withdrawn for investigation
  5. Drainage of the ulcer if there is a collection
  6. Revascularization as needed and indicated by APSV done at visit 0.
  7. Swab from the ulcer for culture and micro-organism count: on detailed visits only.
  8. Debridement as needed.
  9. Dressing:
     * Inspection and assessment of the ulcer
     * Irrigation using 500 ml of saline or as required.
     * Drying of the ulcer (leave to dry)
     * Spread a layer of 3 - 5 mm of Panthenol on a dressing and then apply the dressing to the ulcer
     * Fix the dressing to the ulcer
  Other Names: Panthenol; Ointment; Diabetic foot Ulcer
  Arms: Panthenol

SUMMARY:
Clinical Trial Phase III-b

Study Sponsor:

European Egyptian Pharmaceutical Industries

Sample Size:

120 patients (60 per arm)

Study Population:

Patients with Diabetic foot ulcer of any stage after proper surgical treatment - if needed. Those patients will be recruited from patients attending the Diabetic foot Center at Faculty of Medicine - Alexandria University and the outpatient clinic at Faculty of Medicine, Cairo University.

Recruitment Period: 9 months

Dose application: thick layer of 2-3 mm applied to the dressing then dressing applied to the ulcer.

Endpoints: Complete healing of the ulcer OR 5 months of application of the ointment whichever comes first

DETAILED DESCRIPTION:
Study Design:

This is an open label randomized non-placebo study in which 120 subjects will be randomly allocated to treatment with PedyPhar ointment or Panthenol ointment for their diabetic foot ulcer. Treatment with the ointment will be preceded by appropriate surgical treatment to remove necrotic tissue as indicated by a surgeon for foot ulcer Wagner stages 3-5. Also, diabetic status will be controlled as part of the study. Ointment in either arm will be applied to the ulcer for a maximum of 5 months or till complete healing whichever happens first.

Patients will visit study center every 2 weeks where assessment of the ulcer will be done and patient will be given the ointment for the dressing enough for 2 weeks.

Blood flow in the affected leg will be assessed besides kidney functions complete blood picture besides kidney functions. Diabetic status will be monitored every months and glycosylated hemoglobin will be done every 3 months

Study Duration: 12 months

Study Agent/Intervention Description: PEDYPHAR® is a new patented local ointment composed of natural (Royal Jelly) and (Dexpanthenol) in an innovated, enriched alkaline ointment base.

Dose application: thick layer of 2-3 mm applied to the dressing then dressing applied to the ulcer.

ELIGIBILITY:
Inclusion Criteria:

* Adult diabetic foot syndrome subjects over 18 years of age of any sex
* All stages of diabetic foot syndrome including Wagner stage 5 - Mid-foot gangrene only after appropriate surgical treatment.
* Patients suffering from type 1 or type 2 diabetes mellitus with diabetic foot syndrome.
* Stable metabolic and pharmacological control at recruitment and during the trial period.
* Adequate perfusion of lower limb as measured by HHD and confirmed by APSV.

Exclusion Criteria:

* Non-diabetic foot ulceration (traumatic, thermal ulceration etc)
* Diabetic foot syndrome graded 5 on Wagner's scale - hind foot gangrene only.
* Any pathological state or disease which can affect the development and outcomes of diabetic foot syndrome such as liver cell failure and renal failure
* Severe limb ischemia (by clinical assessment and HHD) unless re-vascularized.
* Presence of slough or sequestrum unless debrided.
* Hemoglobin less than 8 g/dl unless corrected.
* Those receiving NSAIDs, steroids or anti-mitotic drugs.
* Septicemia patients requiring urgent amputation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Healing of the Ulcer | within 5 months or complete healing whichever comes first

SECONDARY OUTCOMES:
reduction of infection in the ulcer site | 5 months
local reaction that may be due to study drug | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Samir H Assaad, PhD, Principal Investigator — Alexandria University Hospitals; Hesham M Abdel Samad, PhD, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Alexandria University Hospitals, Alexandria
  - Cairo University Hospitals, Alexandria

REFERENCES:
- [Derived] Yakoot M, Abdelatif M, Helmy S. Efficacy of a new local limb salvage treatment for limb-threatening diabetic foot wounds - a randomized controlled study. Diabetes Metab Syndr Obes. 2019 Sep 2;12:1659-1665. doi: 10.2147/DMSO.S210680. eCollection 2019. PMID 31564933